CLINICAL TRIAL: NCT06061887
Title: Frequency of Falls in Stroke Patients and Factors Associated With Recurrent Falls
Brief Title: Factors Associated With Recurrent Falls in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Altınay Göksel Karatepe, Professor, Bozyaka Training and Research Hospital
Other Study IDs: 117
Record Dates: First submitted 2023-03-08; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Fall; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fall evaluation — Evaluation of the frequency of falls in patients with acute stroke and determining the risk factors associated with recurrent falls within the first six months after stroke

SUMMARY:
The goal of this observational study is to learn about the recurrent falls in patients with acute stroke. The main question[s] it aims to answer are:

* what is the frequency of recurrent falls
* which factors are associated with recurrent falls in patients with acute stroke.

Participants will be evaluated in terms of

* frequency of recurrent falls within the six months after stroke
* fear of falling
* the stroke severity (Canadian Neurological Scale),
* ambulation level (Functional Ambulation Classification),
* functional disability (Functional Independence Scale)
* Postural control and balance
* functional status (Modified Rankin Scale)

DETAILED DESCRIPTION:
Falling is common in stroke patients both in the hospital and at home after discharge. As a result, physical problems such as fractures and psychological problems such as fear of falling, limitation of physical activity and social isolation occur. Identifying the factors that cause falls after stroke will contribute to the recovery process by preventing complications by taking the necessary precautions and increasing the patient's participation in rehabilitation. This study was planned to determine the frequency of falls in patients with acute stroke and to determine the risk factors associated with recurrent falls within the first six months after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Having an acute stroke over the age of 18
2. To have a cognitive situation to understand and answer questions

Exclusion Criteria:

1. Patients with bilateral hemiplegia
2. Patients without motor involvement
3. Those with a history of stroke
4. Patients with severe cognitive impairment
5. Patients in need of intensive care

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and over, hospitalized in the neurology service with the diagnosis of acute stroke
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Frequency of fall | Six month
  The frequency of recurrent falls were were determined by questioning the patients.

SECONDARY OUTCOMES:
Factors related with recurrent falls | Six month
  Poor postural control, number of falls,fear of falling, functional disability, ambulation level of the patients will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Altınay Göksel Karatepe, MD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences Turkey, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Samuelsson CM, Hansson PO, Persson CU. Determinants of Recurrent Falls Poststroke: A 1-Year Follow-up of the Fall Study of Gothenburg. Arch Phys Med Rehabil. 2020 Sep;101(9):1541-1548. doi: 10.1016/j.apmr.2020.05.010. Epub 2020 Jun 1. PMID 32497600